CLINICAL TRIAL: NCT02584829
Title: Study to Evaluate Cellular Adoptive Immunotherapy Using Polyclonal Autologous CD8+ Antigen-Specific T Cells for Metastatic Merkel Cell Carcinoma in Combination With MHC Class I Up-Regulation and the Anti-PD-L1 Antibody Avelumab
Brief Title: Localized Radiation Therapy or Recombinant Interferon Beta and Avelumab With or Without Cellular Adoptive Immunotherapy in Treating Patients With Metastatic Merkel Cell Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to loss in funding
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: EMD Serono (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Aude Chapuis, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9245; NCI-2014-02462 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHCRC 9245; 9245 (Other: Fred Hutch/University of Washington Cancer Consortium); K24CA139052 (NIH); P30CA015704 (NIH); R01CA176841 (NIH); RG1015013 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2015-10-21; First posted 2015-10-23 (Estimated); Results first posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-02

CONDITIONS: Merkel Cell Polyomavirus Infection; Stage IV Merkel Cell Carcinoma AJCC v7
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — avelumab; Radiotherapy; Radiation; Interferon-beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (avelumab and MHC class I up-regulation) (Experimental): Patients who do not have a HLA type for which T cells can be generated or for whom T cells cannot be generated for technical issues receive avelumab intravenously (IV) over 1 hour every 2 weeks for 12 months. Within 7-10 days after completion of 1-3 doses of avelumab, patients receive MHC class I up-regulation intervention comprising either localized radiation therapy or recombinant interferon beta via intra-tumor injection.
  Interventions: Drug: Avelumab; Other: Laboratory Biomarker Analysis; Radiation: Radiation Therapy; Biological: Recombinant Interferon Beta
- Group 2 (avelumab, MHC class I up-regulation, T cells) (Experimental): Patients who have an HLA type for which T cells can be generated receive avelumab IV over 1 hour every 2 weeks for 12 months. Patients also receive MHC class I up-regulation intervention as in Group 1 between 7-10 days after the first infusion of avelumab and 2-5 days before the first infusion of MCPyV TAg-specific polyclonal autologous CD8+ T cells. Patients receive two infusions of MCPyV TAg-specific polyclonal autologous CD8+ T cells IV over 60-120 minutes.
  Interventions: Drug: Avelumab; Other: Laboratory Biomarker Analysis; Biological: MCPyV TAg-specific Polyclonal Autologous CD8-positive T Cells; Radiation: Radiation Therapy; Biological: Recombinant Interferon Beta

INTERVENTIONS:
Drug: Avelumab — Given IV
  Other Names: Bavencio; MSB-0010718C; MSB0010718C
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: MCPyV TAg-specific Polyclonal Autologous CD8-positive T Cells — Given IV
  Arms: Group 2 (avelumab, MHC class I up-regulation, T cells)
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Biological: Recombinant Interferon Beta — Given via intra-tumor injection
  Other Names: Beta Interferon; Betantrone; Feron; Human Interferon Beta; Interferon Beta; Interferon, Beta; Interferon-B; Interferon-beta; Naferon

SUMMARY:
This phase I/II trial studies the side effects and how well localized radiation therapy or recombinant interferon beta and avelumab with or without cellular adoptive immunotherapy works in treating patients with Merkel cell carcinoma that has spread to other parts of the body. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Interferon beta is a substance that can improve the body's natural response and may interfere with the growth of tumor cells. Monoclonal antibodies, such as avelumab, may help T lymphocytes kill tumor cells. For cellular adoptive immunotherapy, specific white blood cells are collected from the patient's blood and treated in the laboratory to recognize Merkel cell carcinoma. Infusing these cells back into the patient may help the body build an effective immune response to kill Merkel cell carcinoma. Giving localized radiation therapy or recombinant interferon beta and avelumab with or without cellular adoptive immunotherapy may be a better treatment for Merkel cell carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess and compare the safety and potential toxicities associated with treating patients with metastatic Merkel cell carcinoma (MCC) with either major histocompatibility complex (MHC) up regulation and programmed cell death 1 (PD1)-axis blockade (Group 1), or MHC up-regulation, PD1-axis blockade and adoptive transfer of Merkel cell polyoma virus (MCPyV) T antigen (TAg)-specific polyclonal autologous cluster of differentiation (CD)8+ T cells (Group 2).

II. Assess and compare the antitumor efficacy associated with treating patients with metastatic MCC with either MHC up-regulation and PD1-axis blockade (Group 1), or MHC up-regulation, PD1-axis blockade and adoptive transfer of MCPyV TAg-specific polyclonal autologous CD8+ T cells (Group 2).

SECONDARY OBJECTIVES:

I. Examine the in vivo persistence and, where evaluable, migration to tumor sites of adoptively transferred polyclonal CD8+ T cells targeting the MCPyV TAg (Group 2).

II. Examine the in vivo functional capacity of adoptively transferred polyclonal CD8+ T cells targeting the MCPyV Tag (Group 2).

III. Examine and compare evidence of epitope spreading with either MHC up-regulation and adoptive transfer of MHC up-regulation and PD1-axis blockade (Group 1), or MHC up regulation, PD1-axis blockade and adoptive transfer of MCPyV TAg-specific polyclonal autologous CD8+ T cells (Group 2).

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP 1: Patients who do not have a human leukocyte antigen (HLA) type for which T cells can be generated or for whom T cells cannot be generated for technical issues receive avelumab intravenously (IV) over 1 hour every 2 weeks for 12 months. Within 7-10 days after completion of 1-3 doses of avelumab, patients receive MHC class I up-regulation intervention comprising either localized radiation therapy or recombinant interferon beta via intra-tumor injection.

GROUP 2: Patients who have an HLA type for which T cells can be generated receive avelumab IV over 1 hour every 2 weeks for 12 months. Patients also receive MHC class I up-regulation intervention as in Group 1 between 7-10 days after the first infusion of avelumab and 2-5 days before the first infusion of MCPyV TAg-specific polyclonal autologous CD8+ T cells. Patients receive two infusions of MCPyV TAg-specific polyclonal autologous CD8+ T cells IV over 60-120 minutes.

In both groups, MHC class I up-regulation treatment with or without T cell infusions may repeat if indicated.

After completion of study treatment, patients are followed up at 12 months and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Confirmation of MCC by internal pathology review of initial or subsequent biopsy or other pathologic material
* If an accessible lesion is present, a biopsy will be performed within 6 weeks of the start of study intervention; the results of the biopsy must be obtained prior to initiation of study intervention
* Evidence of MCPyV TAg tumor expression by immunohistochemistry on any prior or current tumor specimen or viral oncoprotein antibody confirmation within 6 weeks of the start of study intervention
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 2 at trial entry
* Patients must have at least one bi-dimensionally measurable lesion by palpation, clinical exam, or radiographic imaging within 6 weeks of the start of study intervention (X-ray, computed tomography [CT] scan, positron emission tomography [PET] scan, magnetic resonance imaging [MRI], or ultrasound)
* For patients designated to be treated on Group 2: cardiac ejection fraction >= 35%; for patients with significant risk factors for coronary artery disease (Framingham risk score > 15%), a cardiac stress test is recommended
* At least 3 weeks must have passed since any of the following: systemic corticosteroids, immunotherapy (for example, T-cell infusions, immunomodulatory agents, interleukins, MCC vaccines, intravenous immunoglobulin, expanded polyclonal tumor infiltrating lymphocytes [TIL] or lymphokine-activated killer [LAK] therapy), pentoxifylline, other small molecule or chemotherapy cancer treatment, other investigational agents or other systemic agents that target Merkel cell carcinoma

Exclusion Criteria:

* Known active infections or oral temperature > 38.2 Celsius (C) fewer than 72 hours prior to receiving study treatment or systemic infection requiring chronic maintenance or suppressive therapy
* White blood cells (WBC) < 200/mcl
* Hemoglobin (Hb) < 8 g/dL
* Absolute neutrophil count (ANC) < 1000/mcl
* Platelets < 50,000/mcl
* New York Heart Association functional class III-IV heart failure, symptomatic pericardial effusion, stable or unstable angina, symptoms of coronary artery disease, congestive heart failure, clinically significant hypotension, or history of an ejection fraction of =< 30 % (echocardiogram or multi gated acquisition scan [MUGA])
* Clinically significant pulmonary dysfunction, as determined by medical history and physical exam; patients so identified will undergo pulmonary functions testing and those with forced expiratory volume in 1 second (FEV1) < 2.0 L or diffusion capacity of the lung for carbon monoxide (DLco) (corrected [corr] for hemoglobin [Hgb]) < 50% will be excluded
* Creatinine clearance < 30 ml/min which cannot be attributed to MCC metastasis
* Total bilirubin > 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 2.5 x ULN; for patients with liver metastases: AST/ALT > 5 x ULN
* Active autoimmune disease (e.g. systemic lupus erythematosus, vasculitis, infiltrating lung disease, inflammatory bowel disease) whose possible progression during treatment would be considered unacceptable by the investigators
* Symptomatic and untreated central nervous system (CNS) metastasis; however, patients with 1 to 2 asymptomatic, less than 1 cm brain/CNS metastases without significant edema may be considered for treatment; if sub-centimeter CNS lesions are noted at study entry, then repeat imaging will be performed, if more than 4 weeks have elapsed from the last scan
* Any condition or organ toxicity that is deemed by the principal investigator (PI) or the attending physician to place the patient at unacceptable risk for treatment on the protocol
* Pregnant women, nursing mothers, men or women of reproductive ability who are unwilling to use effective contraception or abstinence; women of childbearing potential must have a negative pregnancy test within 2-6 weeks prior to treatment
* Clinically significant and ongoing immune suppression including, but not limited to, systemic immunosuppressive agents such as cyclosporine or corticosteroids, chronic lymphocytic leukemia (CLL), uncontrolled human immunodeficiency virus (HIV) infection, or solid organ transplantation
* Patients may not be on any other treatments for their cancer aside from those included in the protocol; patients may not undergo another form of treatment concurrently with this study
* Known severe hypersensitivity reactions to monoclonal antibodies (grade >= 3 National Cancer Institute [NCI]-Common Terminology Criteria for Adverse Events [CTCAE] version [v] 4.0), any history of anaphylaxis, or uncontrolled asthma
* Vaccination with live inactivated viral strains for the prevention of infectious diseases within 4 weeks of the start of the study treatment, inactivated influenza vaccines are permitted while on trial
* Known alcohol or drug abuse
* Legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aude Chapuis, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 (Avelumab and MHC Class I Up-regulation) | Group 2 (Avelumab, MHC Class I Up-regulation, T Cells)
Started | 1 | 7
Completed | 0 | 3
Not Completed | 1 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Progressive Disease | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Avelumab and MHC Class I Up-regulation) | Group 2 (Avelumab, MHC Class I Up-regulation, T Cells) | Total
Number analyzed (Participants) | 1 | 7 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 7 | 7
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 1 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 7 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 7 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 7 | 8

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Response, Based on Median Time to New Metastasis
Description: Median time to new metastases reported for each group below. Group 1 result is NA, patient had no new detectable metastases in study follow-up period. Arm I is not analyzed because the one patient in Arm I did not experience new metastasis in their followup period, so they are not evaluable.
Time Frame: Up to 1 year
Population: Patient in group 1 did not experience new metastasis in followup period of 1 year. Only 4 patients in group 2 experienced new metastases in the followup period of 1 year. The other 3 patients in group 2 were omitted due to no new metastases.
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Group 2 (Avelumab, MHC Class I Up-regulation, T Cells)
Number analyzed (Participants) | 4
Days | 53 (23.45)

2. Primary Outcome: Count of Participants Who Experienced Adverse Events, Evaluated According to the Current Guidelines in National Cancer Institute (NCI) Common Toxicity Criteria Version 4.0
Description: Evidence and nature of toxicity related to the treatment will be assessed and compared between groups.
Time Frame: Up to 4 weeks after the last infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Avelumab and MHC Class I Up-regulation) | Group 2 (Avelumab, MHC Class I Up-regulation, T Cells)
Number analyzed (Participants) | 1 | 7
Participants | 1 | 6

3. Secondary Outcome: Disease Response, as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1
Description: Patients were evaluated for their disease response throughout their follow up period. Disease response reported is best response per patient. A complete response (CR) will be defined as total regression of all tumors, a PR as 30% or greater decrease in the sum of the longest diameter of target lesions compared to baseline and PD as 20% increase in the sum of the longest diameter of target lesions compared to the smallest prior diameter (RECIST v1.1 criteria).
Time Frame: 28 days post infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Avelumab and MHC Class I Up-regulation) | Group 2 (Avelumab, MHC Class I Up-regulation, T Cells)
Number analyzed (Participants) | 1 | 7
Participants
  Complete Response | 1 | 2
  Partial Response | 0 | 1
  Stable Disease | 0 | 0
  Progressive Disease | 0 | 3
  Partial Complete Response | 0 | 1

4. Secondary Outcome: Count of Participants That Displayed Evidence of Epitope Spreading
Description: Quantiﬁcation of the overall recognition of the MCPyV T-antigen for each patient will likely be performed by testing the reactivity of whole peripheral blood mononuclear cells (PBMC) before and at indicated timepoints after treatment to peptides 15 amino acids (aa) in length offset by 5 aa bases spanning the whole T-antigen protein to include both CD8 and CD4 responses regardless of the HLA type of the patient. Due to changes in assay technology, epitope spreading was detected using a flow cytometric based intracellular cytokine assay.
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2 (Avelumab, MHC Class I Up-regulation, T Cells)
Number analyzed (Participants) | 7
Participants | 2

5. Secondary Outcome: Functional Capacity of Transferred T Cells (Group 2)
Description: To evaluate the direct ex vivo function of the transferred cells, where possible, tetramer+ cells within collected peripheral blood mononuclear cells (PBMCs) will be evaluated for production of intracellular cytokines including interferon (IFN), tumor necrosis factor alpha and interleukin-2 in response to cognate antigen using an intracellular cytokine assay. This endpoint was evaluable in 4 of 7 patients, all 4 of whom upregulated interferon, tumor necrosis factor alpha and IL-2 expression in response to cognate antigen using intracellular cytokine assay. Persistence was not detected for 3 out of 7 patients in group 2, making them unevaluable for functional capacity.
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2 (Avelumab, MHC Class I Up-regulation, T Cells)
Number analyzed (Participants) | 4
Participants | 4

6. Secondary Outcome: Merkel Cell Carcinoma (MCC)-Specific Survival
Description: Survival status in patients with Merkel cell carcinoma will be evaluated. Data is reported as count of participants that survived past the 1 year follow up period.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Avelumab and MHC Class I Up-regulation) | Group 2 (Avelumab, MHC Class I Up-regulation, T Cells)
Number analyzed (Participants) | 1 | 7
Participants | 1 | 6

7. Secondary Outcome: Count of Participants Who Displayed Persistence of Transferred T Cells in Blood and Tumor (Group Co2)
Description: Persistence of trasferred T cells was evaluated and assessed after 90 days. Patients were counted if transferred T cells were detected beyond 90 days.
Time Frame: Up to 90 days post infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2 (Avelumab, MHC Class I Up-regulation, T Cells)
Number analyzed (Participants) | 7
Participants | 4

ADVERSE EVENTS:
Time Frame: Up to 12 months after infusion
Description: All unexpected and serious AEs which may be due to study treatment or intervention must be reported to the FHCRC Institutional Review Office (IRO) per their current reporting requirements.
  All grade ≥ 3 CTCAE v.4 AEs will be collected through 4 weeks after each participant's last T-cell infusion and per section 12.C. Beginning 4 weeks after the participant's last infusion, only study related toxicities will be collected.ci
Arm/Group | Group 1 (Avelumab and MHC Class I Up-regulation) | Group 2 (Avelumab, MHC Class I Up-regulation, T Cells)
All-Cause Mortality (participants affected / at risk) | 0/1 | 3/7
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/7
Other Adverse Events (participants affected / at risk) | 1/1 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Avelumab and MHC Class I Up-regulation) (N=1) | Group 2 (Avelumab, MHC Class I Up-regulation, T Cells) (N=7)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Avelumab and MHC Class I Up-regulation) (N=1) | Group 2 (Avelumab, MHC Class I Up-regulation, T Cells) (N=7)
Lymphocyte count decreased (Investigations) | 1 (1) | 4 (8)
Fever (General disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT02584829/Prot_SAP_000.pdf